CLINICAL TRIAL: NCT06998290
Title: Feasibility of Home Telemonitoring of Infants With Congenital Heart Disease Awaiting Surgery During the First Year of Life: the Blue-Line Pilot Study
Brief Title: Feasibility of Home Telemonitoring of Infants With Congenital Heart Disease Awaiting Surgery During the First Year of Life
Acronym: Blue-Line
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2021/41; 2024-A01759-38 (Other: ID-RCB number)
Record Dates: First submitted 2025-03-18; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: CHD - Congenital Heart Disease
Keywords: Congenital heart disease; Infants; Vulnerability; Home monitoring; Therapeutic education; Digital platform
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blue-Line programme (Experimental): Telemonitoring program
  Interventions: Other: Blue-Line home telemonitoring program

INTERVENTIONS:
Other: Blue-Line home telemonitoring program — * A dedicated telemonitoring team with nurses and pediatric cardiologist
  * A dedicated therapeutic patient education programme
  * A home telemonitoring medical device with a dedicated platform

SUMMARY:
Actually, there is no telemonitoring program that includes newborns or infants with congenital heart disease awaiting cardiac intervention. This is a vulnerable period, prone to clinical complications, rehospitalization, parental stress, and requires monitoring with clinical and therapeutic optimization. The aim of the study is to assess the feasibility and acceptability of monitoring newborns and infants with congenital heart disease awaiting cardiac surgery using the Blue-Line home telemonitoring program.

DETAILED DESCRIPTION:
Today, congenital heart disease affects around 0.8% of births in France. One third of children diagnosed antenatally or postnatally with congenital heart disease will require surgical or percutaneous intervention within the first year of life. Actually, there is no telemonitoring program that includes newborns or infants with congenital heart disease awaiting cardiac intervention. This is a vulnerable period, prone to clinical complications, rehospitalization, parental stress, and requires monitoring with clinical and therapeutic optimization. Our research team at the M3C Network Reference Center aims to develop home telemonitoring for these patients, in order to innovate and optimize their care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and/or infants aged 0 to 12 months inclusive at the time of diagnosis.
* With congenital heart disease as defined in the ICD-11 classification.
* Waiting for an intervention by cardiac surgery or interventional catheterization.
* Free, informed consent signed by the holder(s) of parental authority.
* Person affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Short-term vital prognosis
* Clinical situation identified at the M3C RCP that contraindicates a return home
* Family situation identified at the M3C RCP as contra-indicating a return home
* Extra-cardiac co-morbidities requiring hospitalisation independent of the heart disease (e.g. severe renal failure, neurological deficit, complex immune deficiency, etc.).
* Limited understanding of parental authority holder(s) / caregivers (non-French speaking, hearing impaired, cognitive impairment or other)
* Parents unable to give informed consent.
* Minors with parental authority

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the implementation of the patient therapeutic education programme: number of validated workshops out of number of workshops offered | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Evaluation of the measurement devices: functional (yes/no) | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Evaluation of the telemonitoring platform (functional/ergonomic/reliable) | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Recruitment rate: number of participants out of number of eligible patients | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Adherence to the telemonitoring programme: number of the participants who finish the programm out of number of patients included | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Acceptability to parents: parent satisfaction questionnaire | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria
Acceptability to caregivers: caregiver satisfaction questionnaire | between inclusion visit and the last protocol visit (month 12)
  Contributes to programme feasibility criteria

SECONDARY OUTCOMES:
Events of interest | between months 3 and 12
  Events of interest are defined as any event leading to discontinuation of remote monitoring and/or unscheduled hospitalisation.
Date of telemonitoring alert | between months 3 and 12
  Contributes to the alert performance criteria
Severity level of alert (orange/red) | between months 3 and 12
  Contributes to the alert performance criteria
Appropriateness of the alert (yes/no) | between months 3 and 12
  Contributes to the alert performance criteria
Respect for the procedure to be followed following an alert by parents (yes/no) | between months 3 and 12
  Contributes to the alert performance criteria
Appropriateness of medical management following the alert given the clinical situation (yes/no) | between months 3 and 12
  Contributes to the alert performance criteria
Evolution of the height (cm) | between months 2 and 12
  Contributes to the clinical evolution criteria
Evolution of the weight (kg) | between months 2 and 12
  Contributes to the clinical evolution criteria
Evolution of oxygen saturation (SpO2, %) | between months 2 and 12
  Contributes to the clinical evolution criteria
Evolution of the heart failure score (Ross classification) | between months 2 and 12
  Contributes to the clinical evolution criteria
Life quality | between months 2 and 12
  Changes in the score of the QUALIN (QUALIté de vie du Nourrisson) validated generic quality of life proxy questionnaire: before returning home, at 3 months and at the end of the programme. The QUALIN questionnaire is a 34-item generic French QoL instrument designed for infants (aged 0-3 years). Each answer scores from -2 (totally false) to +2 (quite true). An item with a score >1 corresponds to favourable QoL.
Parental anxiety | between months 2 and 12
  Changes in the score of the STAI (State-Trait Anwiety Inventory) parental anxiety questionnaire: state-trait anxiety inventory. The STAI questionnaire is a 40-item instrument designed for adults. Each answer score from 1 to 4. The higher the score, the less anxious the patient.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier, France
  - CHU de Bordeaux - Hôpital Cardiologique Haut Lévêque, Pessac, France